CLINICAL TRIAL: NCT06059105
Title: Immediate Implant Using an Inverted Co-Axis at 12º Versus a Conventional Conical Implant: A Randomised Clinical Trial With 1 Year Follow-up
Brief Title: Immediate Implant Using an Inverted Co-Axis at 12º Versus a Conventional Conical Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, JAVIER GAMON, Clinical Project Manager Dentistry faculty, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIR-ELC-2021-09
Record Dates: First submitted 2023-09-04; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dental Implant Failed
Keywords: co-axis implant; dental implant; implant angulation; success rate; marginal bone loss

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into two groups. The test group (n=15) will be treated with the Inverta Co-Axis 12º implant (Southern Implants). In the control group (n=15) the Internal Conical implants (Southern implants) will be used. The difference between both implants lies in the fact that the Inverta Co-Axis 12º implant presents two different variants to the classic implant with parallel walls (Internal Conical)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Inverted Co-Axis 12º Southern Implants (15 patients): The implant is placed in the center of the socket due to that has an angled neck of 12º, which allows the implant to be placed in the center of the alveolus, optimizing the alveolar bone and improving the prosthetic emergence. This is due to the access of the screw being located palatally, simplifying the restoration of the crown, avoiding cemented crowns, lowering the laboratory cost and of prosthetic accessories.
  Interventions: Device: Immediate Implant Surgery
- Control Group (Active Comparator): Internal Conical (Deep Tapered Conical) South Implants (15 patients): conventional conical implant with internal connection. The implant is placed palatally in order to have a good emergence profile.
  Interventions: Device: Immediate Implant Surgery

INTERVENTIONS:
Device: Immediate Implant Surgery — Inverted Co-Axis 12º Southern Implants
  Arms: Test Group
Device: Immediate Implant Surgery — Internal Conical (Deep Tapered Conical) South Implants
  Arms: Control Group

SUMMARY:
This study is a randomised controlled clinical trial. The patients will be included for the placement of immediate implants with immediate crown placement, to replace maxillary anterior teeth. Any significant differences between the Co-Axis implant and a conventional conical implant will be evaluated.

DETAILED DESCRIPTION:
Introduction: It is commonly known that the placement of an immediate implant is a technique-sensitive procedure, as the implant should be placed in the palatal aspect for the perfect prosthetic emergence and profile. In order to supply this complexity, there is a novel macroimplant design involving an implant with a 12º angled platform. This angulation of the coronal part of the implant allows perfect emergence of the placement of post-extraction implants, since it is placed at the center of the socket, acquiring the best possible bone. In addition, thanks to the angled neck, prosthetic emergence is ideal, as it is corrected and emerges through the cingulate area, thus securing a perfect emergence profile.

Objectives:

Primary Outcomes: Evaluate the percentage of success and survival of the Inverted Co-Axis 12º Southern Implants versus the Internal Conical (Deep Tapered Conical) South Implants on a 1-2-1 follow-up.

Secondary Outcomes:

1. To evaluate the primary stability of both implant systems through a coefficient stability if implants using the Penguin RFA;
2. To evaluate the horizontal and vertical marginal bone loss via a CBCT, 1 year after implant placement;
3. To evaluate the soft tissues via the Pink Esthetic Score (PES) 1 year post-op.

Materials and Methods: Patients were randomly assigned in 2 groups of 15 patients, conical or inverta co-axis implants. Immediate implants in the aesthetic zone of the superior maxilar were placed with an immediate provisional crown restoration. In the same surgery, a connective tissue graft was performed. Only type I sockets according to the Elian Classification were eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented with a good well-being status and no contraindication for undergoing an oral surgical procedure
* Patients aged 18 and over
* Adequate oral hygiene, with patient's presenting a plaque index lower than 15% using the Index Scale publish by Löe et al.
* Patients who demonstrated motivation and compiled by attending the allocated follow-up appointments
* One single tooth indicated to be extracted due to having a poor prognosis in the maxilla (central or lateral incisors, canines or premolars)
* Absence of vestibular dehiscence in the bone table and presence of soft tissue without recession (Alveolus type I according to the classification of Elian et al. which could be determined on the day of surgery
* Sufficient bone to allow implant placement with primary stability
* To avoid image blurring or artefacts during CBCT, patients were included if they did not have a bridge or amalgam restoration close to the implant placement.

Exclusion Criteria:

* If the patient presented with an acute infection in the tooth where the implant is to be placed
* Absence of posterior sector in which it would cause an occlusal overload
* Alveolus with enough space to place an implant with a diameter of 4.5mm (since implants with a 3.5 coronal diameter have a widening in the middle third of the implant of 4.5mm)
* Patients with an unstable periodontal status
* Patients who smoked more than 10 cigarettes a day
* Patients who had medical histories which contraindicate implant surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 1 year
  ICOI Pisa Implant quality of Health Criteria
Survival Rate | 1 year
  "the implant is still in mouth",

SECONDARY OUTCOMES:
Horizontal and Vertical bone Changes | 1 year
  Three CBCT will be made (CBCT 1- before implant placement, CBCT 2- just after implant placement, CBCT 3- 1 year before implant placement). First year bone loss overlap CBCT 1, 2 and 3. The horizontal bone changes will be from the implant platform at 1, 3 and 5mm from it. The vertical measurements will be from implant platform till the most vestibular and palatal bone peak.
Implant primary stability | Right after the implant placement
  Recorded using Penguin RFA device
Status of the soft tissues | At 1 year
  The Pink Esthetic Score (PES) is based on seven variables: mesial papilla, distal papilla, soft tissue contour, gingival margin level, alveolar process deficiency, soft tissue colour and texture. Each variable will be evaluated with a score of 2-1-0, with 2 being the best score and 0 the worst score. The maximum score, which reflects a perfect coincidence of the peri-implant soft tissue with that of the reference tooth, is 14.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain